CLINICAL TRIAL: NCT01941043
Title: A Randomized, Double-Blind, Placebo-Controlled, Sequential Parallel Study of CERC-301 in the Adjunctive Treatment of Subjects With Severe Depression and Recent Active Suicidal Ideation Despite Antidepressant Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avalo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Clin301-201
Record Dates: First submitted 2013-09-05; First posted 2013-09-13 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-12

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- CERC-301, Treatment Sequence 1 (Experimental): Treatment Sequence 1 - 7 days on placebo and 28 days on study drug (either 12mg or 8mg)
  Interventions: Drug: CERC-301; Other: Placebo
- CERC-301, Treatment Sequence 2 (Experimental): Treatment Sequence 2 - Placebo for 7 days and study drug for 28 days (8 mgs)
  Interventions: Drug: CERC-301; Other: Placebo
- Placebo, Treatment Sequence 3 (Placebo Comparator): Treatment Sequence 3 - Placebo for 35 Day treatment period
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CERC-301
  Arms: CERC-301, Treatment Sequence 1; CERC-301, Treatment Sequence 2
Other: Placebo

SUMMARY:
The current study will evaluate the antidepressant effect of CERC-301 during 28 days of treatment in subjects with MDD who are currently experiencing a severe depressive episode despite stable ongoing treatment with selective serotonin- or serotonin-norepinephrine reuptake inhibitors (SSRI or SNRI). The study population will be enriched for subjects that would benefit most from rapid onset, those with recent active suicidal ideation, but not a risk to themselves or others and are deemed appropriate for an out-patient study with careful safety surveillance. This will allow the study to focus on the antidepressant effects of CERC-301 but also explore effects on suicidal ideation. To explore rapid onset, the primary endpoint will be at 7 days, but effects over the 28 days of treatment will be examined as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 70 years of age inclusive.
2. Females must be either:

   1. Post-menopausal (amenorrhea for at least 12 consecutive months), surgically sterile -or-
   2. Women of childbearing potential (WOCBP) meeting the criteria below:

   i. Uses an acceptable double-barrier method of contraception as determined by the Investigator -and- ii. Is not lactating, has a negative serum beta human chorionic gonadotropin pregnancy test at screening and a negative urine pregnancy test prior to randomization on Day 0.
3. Male subjects must agree to use a condom if partner is of childbearing potential.
4. Diagnosis of MDD recurrent without psychotic features according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria with diagnosis confirmed using the Structured Clinical Interview for DSM-IV Axis I Disorders Clinical Trials Version (SCID-CT).
5. Currently adhering to antidepressant drug regimen that consists of stable SSRI or SNRI therapy
6. Inadequate antidepressant response to current antidepressant therapy despite adequate dose and duration
7. HDRS-17 score ≥ 21 on the HDRS-17 performed by the site at screening
8. Recent active suicidal ideation defined as a score of 2 on the intensity of ideation section on the Columbia-Suicide Severity Rating Scale (C-SSRS) during the four weeks prior to screening using the "Baseline/Screening" version of the C-SSRS.
9. In otherwise good general health without any unstable medical conditions (as determined by medical history, physical examination, 12-lead ECG, clinical laboratory testing, etc.).

Exclusion Criteria:

1. History of substance abuse or dependence within the 3 months prior to screening.
2. Positive urine drug test at screening and prior to randomization on Day 0 unless due to a permitted medication that is documented in the subject's medication history.
3. Positive ethanol breath test at screening and/or prior to randomization on Day 0.
4. Elevated semi-recumbent blood pressure at screening and prior to randomization on Day 0, defined as systolic blood pressure > 140 mm Hg and diastolic blood pressure
5. Active, comorbid disease that might limit the ability of the subject to participate in the study as determined by the Investigator (i.e. poorly controlled diabetes mellitus, unstable angina, coronary artery disease, congestive heart failure, etc.).
6. Subjects with clinical laboratory test abnormality deemed clinically significant by the Investigator at screening.
7. Axis I diagnosis of obsessive compulsive disorder, posttraumatic stress disorder, bipolar I or II mood disorders, eating disorders (e.g., anorexia nervosa, bulimia nervosa), psychotic disorders (e.g., schizoaffective disorder, schizophrenia), significant cognitive disorders (e.g., delirium, dementia, amnesia), or dissociative disorders.
8. Subjects with Axis II diagnosis of borderline, antisocial, paranoid, schizoid, schizotypal, or histrionic personality disorder.
9. Subjects with a neurologic disorder that could cause or contribute to depression (e.g., Alzheimer's disease, Parkinson's disease).
10. Female subjects currently experiencing postpartum depression.
11. Subjects who, in the opinion of the Investigator, are not appropriate for a 35-day placebo-controlled study due to risk of significant threat to self or others during screening or study conduct.
12. Use of other NMDA-receptor modulators (e.g., dextromethorphan, ketamine, amantadine, memantine) within 30 days of screening and throughout the study.
13. The following concomitant medication use is excluded within six weeks prior to screening:

    * Bupropion or tricyclic antidepressants
    * Intermittent, symptomatic use of benzodiazepines (e.g. symptomatic treatment of anxiety or panic attacks)
    * Antipsychotics
    * Lithium
    * Any medications known to directly interact with central or peripheral serotonergic receptors, other than the permitted antidepressants.
    * Any medications known to directly interact with central noradrenergic receptors, other than the permitted antidepressants.
14. Electroconvulsive therapy, transcranial magnetic stimulation, or vagal nerve stimulation during the current depressive episode.
15. Participation in an investigational drug or device study within the 6 months prior to screening.
16. Subjects with suicidal behavior within 6 months prior to screening as measured by the C-SSRS "Baseline/Screening" version.
17. Subjects with a C-SSRS score > 2 on the intensity of ideation section at randomization (Visit 2a), using the "Since Last Visit" version of the C-SSRS.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1357 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
HDRS-17 after 7 days of dosing with study drug | Screening & Days 0, 4, 7, 11, 14, 21,28, & 35
  The overall between-treatment difference will be computed as the weighted average of the differences (drug vs. placebo)

SECONDARY OUTCOMES:
HDRS-17 Averaged between 7 and 28 days of treatment with study drug | Screening, Days 0, 4, 7, 11, 14, 21, 28, & 35
  This will be analyzed using the mixed effects model for repeated measures. The between-group (drug vs. placebo) differences will be estimated by the least squares mean for the contrast in the main effect.
HDRS-17 after 28 days of dosing with study drug | Screening, Days 0, 4, 7, 11, 14, 21, 28, 35
  This will be analyzed using the mixed effects model for repeated measures . The between-group difference will be estimates by the least squares mean difference at Day 28 as a simple contrast from the model.

CONTACTS AND LOCATIONS:
Overall Officials: James Vornov, MD, PhD, Study Director — Avalo Therapeutics, Inc.
Locations (24):
- United States (24):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona TMS Therapy Center, Phoenix, Arizona
  - ProScience Research Group, Culver City, California
  - Collaborative NeuroScience Network, Inc., Garden Grove, California
  - Behavioral Research Specialists, Glendale, California
  - Synergy Clinical Research Center, National City, California
  - Pacific Clinical Trials, LLC, Oakland, California
  - Southern CA Psychiatrists, Oceanside, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Clinical Neuroscience Solutions, Jacksonville, Florida
  - Scientific Clinical Research, Inc., North Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Chicago Psychiatry Associates, Chicago, Illinois
  - Sheppard Pratt Health System, Baltimore, Maryland
  - PCRC, O'Fallon, Missouri
  - Bioscience Research, Mount Kisco, New York
  - The Medical Research Network, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Northwest Clinical Research Center, Bellevue, Washington